CLINICAL TRIAL: NCT02105571
Title: Social Support During a Randomized Trial of a Trucker Weight Loss Intervention
Brief Title: Evaluation of Safety and Health Involvement For Truck Drivers
Acronym: SHIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Olson, Scientist, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: e3061; R01HL105495 (NIH)
Record Dates: First submitted 2014-02-28; First posted 2014-04-07 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Body Weight; Nutrition; Physical Activity; Sleep; Health Promotion; Stress; Safety
MeSH Terms: conditions — Obesity; Body Weight; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention activities take place over a 6-month period for each participant, and include a weight loss competition with self-monitoring and feedback; computer-based training units on healthy weight loss, healthy eating, exercise, and sleep; and up to four motivational interviews with a health coach by cell phone.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Continued work conditions and "Usual Practices" in that workplace

INTERVENTIONS:
Behavioral: Intervention
  Arms: Intervention

SUMMARY:
The current project is a randomized, controlled evaluation of a new weight loss and health promotion intervention for truck drivers. The intervention is a 6-month weight loss competition supported with computer based training, behavioral self-monitoring, and motivational interviewing. We hypothesize that the intervention will produce greater change than a usual practices control condition. Our secondary hypothesis is that social support and stress in home and work environments will moderate intervention efficacy.

DETAILED DESCRIPTION:
Commercial truck drivers have overweight and obesity rates that may be 20% higher than the general population. Obesity has established mortality and disease consequences, including heart disease, diabetes, and sleep apnea. Driver health is also an important safety hazard because obesity and sleep apnea increase the risk of crashes. Drivers experience multiple roadblocks to health, including an isolating job structure that restricts physical activity and dietary choices. Despite the growing health crisis, there is a lack of effective weight loss and health promotion interventions for truck drivers. We therefore developed an intervention that is integrated with the job structure and modern technologies of truck driving. The intervention is a 6-month weight loss competition supported with computer based training, behavioral self-monitoring, and motivational interviewing. The study is a cluster randomized trial where worksites (terminals) will be randomized to intervention and control conditions. We will collect measures from drivers at baseline (month 0), post-intervention (month 6), and one-year follow-up (month 18). The project will take place over five years and accomplish three specific aims:

1. Determine intervention efficacy for producing changes in diet, exercise, and body weight. Previous weight loss interventions for truck drivers have been minimally effective, and there is a need to evaluate new approaches with randomized, controlled designs. Therefore, we will randomize matched pairs of worksites (terminals) to intervention and control conditions. Drivers at intervention terminals will complete intervention activities over a 6-month period. Drivers at control terminals will receive no treatment during the same time period. Primary outcomes will be changes in body weight, fruit and vegetable consumption, high-saturated fat and high-sugar food consumption, and physical activity.
2. Determine whether baseline social support and stress moderate intervention efficacy. Although social support and stress have established effects on weight loss with other populations, we know little about the role of social support and stress during interventions for truck drivers. Therefore, we will measure social support and stress in home and work environments at each measurement time point. After the intervention, and again at one-year follow-up, we will test whether social support and stress factors moderated subsequent behavior change and weight loss.
3. Measure the integrity of each intervention component and model how the intervention worked. We are evaluating a new multi-component intervention with an understudied population. In order to understand how the intervention worked and guide future research, we will measure fidelity and participation in each intervention component and use mediation analyses to determine how the different components affected study outcomes. Analyses will provide an explicit check of the intervention's theoretical underpinnings and assess whether proposed change processes were achieved.

Accomplishing our aims will significantly advance weight loss and health promotion knowledge to the benefit of over 3 million truck drivers in the US, and potentially generalize to 15 million additional workers who spend substantial time alone or traveling for work.

ELIGIBILITY:
Inclusion Criteria:

* Truck driver currently employed at a participating company
* BMI > 27.0

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body weight at 6 and 18 months | Baseline, 6 months, 18 months
  Directly measured body weight, as well as calculated body mass index based on directly measured height and weight
Change from baseline in dietary behaviors at 6 and 18 months | Baseline, 6 months, 18 months
  Survey measures of: fruit and vegetable intake; calories from fat; sugary food and drink consumption; fast food consumption
Change from baseline in physical activity at 6 and 18 months | Baseline, 6 months, 18 months
  Survey and actigraphy measures of physical activity

SECONDARY OUTCOMES:
Change from baseline in blood pressure at 6 and 18 months | Baseline, 6 months, 18 months
  Direct measurement
Change from baseline in percent body fat at 6 and 18 months | Baseline, 6 months, 18 months
  Direct measurement via Bioelectric Impedance Analysis
Change from baseline in blood lipids and lipoproteins at 6 and 18 months | Baseline, 6 months, 18 months
  Direct measurement of total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides via Cholestech LDX Analyzer
Change from baseline in blood glucose at 6 and 18 months | Baseline, 6 months, 18 months
  Direct measurement via Cholestech LDX Analyzer
Change from baseline in sleep and fatigue at 6 and 18 months | Baseline, 6 months, 18 months
  Psychomotor Vigilance Task; survey measures of: sleep quality; sleep adequacy; sleep apnea risk
Change from baseline in anthropometric measurements at 6 and 18 months | Baseline, 6 months, 18 months
  Direct measurement of waist-to-hip ratio and neck circumference
Change from baseline in stress at 6 and 18 months | Baseline, 6 months, 18 months
  Survey measures of: job stress; general life stress; major life events; work-to-family and family-to-work conflict
Change from baseline in social support at 6 and 18 months | Baseline, 6 months, 18 months
  Survey measures of: social support for diet and exercise from family, friends, coworkers, and others; supervisor support
Change from baseline in self-efficacy at 6 and 18 months | Baseline, 6 months, 18 months
  Self-efficacy for diet and exercise behaviors
Change from baseline in strength and fitness at 6 and 18 months | Baseline, 6 months, 18 months
  Grip strength; 6-minute walk test; hamstring flexibility
Change from baseline in safety outcomes (injuries, crashes, moving violations) at 6 and 18 months | Baseline, 6 months, 18 months
  Survey measures of injuries, crashes, and moving violations; company records of lost-time injuries, crashes, and moving violations
Change from baseline in driving measures (sudden decelerations, driving over the speed limit, fuel efficiency, safety belt use) at 6 and 18 months | Baseline, 6 months, 18 months
  Survey measures of sudden vehicle decelerations, driving over the speed limit, and safety belt use; Engine computer records of sudden vehicle decelerations, driving over the speed limit, and fuel efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Olson R, Anger WK, Elliot DL, Wipfli B, Gray M. A new health promotion model for lone workers: results of the Safety & Health Involvement For Truckers (SHIFT) pilot study. J Occup Environ Med. 2009 Nov;51(11):1233-46. doi: 10.1097/JOM.0b013e3181c1dc7a. PMID 19858740
- [Background] Wipfli B, Olson R, Koren M. Weight-loss maintenance among SHIFT pilot study participants 30-months after intervention. J Occup Environ Med. 2013 Jan;55(1):1-3. doi: 10.1097/JOM.0b013e31827db848. No abstract available. PMID 23291953
- [Derived] Olson R, Wipfli B, Hanson GC, Bodner T, Anger WK, Elliot DL, Mansfield L. Weight loss maintenance among truck drivers in the SHIFT randomised controlled trial, USA. Occup Environ Med. 2025 Jul 9;82(4):168-175. doi: 10.1136/oemed-2024-109903. PMID 40355262
- See also: Related Info — https://www.ohsushift.com